CLINICAL TRIAL: NCT01388972
Title: Assessment of Food Environment and Physical Activity Opportunities in Three Neighbourhoods of Buenos Aires City
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 1656
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Nutrition; Physical Activity
Keywords: Community nutritional environment; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Several environmental factors have contributed to the growing pandemic of obesity. It has been described that some characteristics of food and built environment have an influence on patterns of food consumption and physical activity of people in a certain place.

We have designed a cross-sectional study to describe some aspects of the food environment (community and consumer) and the frequency, distribution and characteristics of the space available to perform physical activity in three neighborhoods of Buenos Aires city.

Three neighborhoods of Buenos Aires (with representativity), from different socioeconomic strata, will be selected by convenience to conduct this study.

The study will consist on three stages: first, the generation of the sampling frame of food stores, public and private spaces available for carrying out physical activity, and the development of a tool designed to evaluate the availability of healthy foods in supermarkets and grocery stores. Finally, a sample of those stores will be randomly selected for assessing the availability of selected foods.

In Argentina, the knowledge of the food environment is limited. We believe that the information obtained in this study will contribute to a better understanding of the subject.

ELIGIBILITY:
Inclusion Criteria:

* Stable Places and ambulant stands (only those that are located habitually in the same place) of food sale and / or drinks of any type.
* Public or private spaces destined for the accomplishment of physical activity.

Exclusion Criteria:

* Places and stands of food sale and / or drinks and spaces for the accomplishment of physical activity not opened the public in general (as those who are inside schools, places of work, centers of health, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A community sample of Recoleta, Almagro and Constitucion neighborhoods of Buenos Aires, Argentina has been conveniently selected by major representation of different socioeconomic stratus. The value of the square meter of the property (2 rooms apartments) was used as indirect indicator of socioeconomic level.
Sampling Method: Probability Sample
Enrollment: 2924 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina